CLINICAL TRIAL: NCT06648031
Title: A Phase 1B, Randomized, Open-label, Active-controlled, Parallel, Multiple-dose Study Comparing the Safety, Pharmacokinetics and Efficacy of Dehydratech Cannabidiol and Glucagon-like Peptide 1 Agonists Alone and in Combination, in Overweight or Obese, pre-and Type 2 Diabetic Participants.
Brief Title: Comparison of the Safety, Efficacy and Pharmacokinetics of DehydraTECH -CBD and DehydraTECH-GLP1 Agonists Alone or in Combination, in Overweight or Obese, Pre- and Type 2 Diabetic Participants
Acronym: DehydraTECH
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Lexaria Bioscience Corp. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GLP-1-H24-4
Record Dates: First submitted 2024-10-16; First posted 2024-10-18 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Type2diabetes
MeSH Terms: interventions — semaglutide; Single Person

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Arm 1 - DehydraTECH-CBD alone (Experimental)
  Interventions: Drug: Arm 1 - DehydraTECH-CBD alone
- Arm 2 - DehydraTECH-semaglutide alone (Experimental)
  Interventions: Drug: Arm 2 - DehydraTECH-semaglutide alone
- Arm 3 - DehydraTECH-CBD in combination with DehydraTECH-semaglutide (Experimental)
  Interventions: Drug: Arm 3 - DehydraTECH-CBD in combination with DehydraTECH-semaglutide
- Arm 4 - Rybelsus medication (semaglutide) alone as a positive control. (Active Comparator)
  Interventions: Drug: Arm 4 - Rybelsus medication (semaglutide) alone
- Arm 5- DehydraTECH Tirzepatide (Experimental)
  Interventions: Drug: Arm 5- Tirzepatide

INTERVENTIONS:
Drug: Arm 1 - DehydraTECH-CBD alone — Dose: 250 mg CBD twice daily (500 mg/day) for 12 weeks. Route of administration: Oral Dosage form: Capsule
  Arms: Arm 1 - DehydraTECH-CBD alone
Drug: Arm 2 - DehydraTECH-semaglutide alone — Dose: 3.5 mg once daily for 4 weeks, ascending to 7 mg once daily for the remaining 8 weeks. Route of administration: Oral Dosage form: Capsule
  Arms: Arm 2 - DehydraTECH-semaglutide alone
Drug: Arm 3 - DehydraTECH-CBD in combination with DehydraTECH-semaglutide — DehydraTECH-CBD dosing = 250 mg twice daily for 12 weeks.
  - DehydraTECH-semaglutide = 3.5 mg once daily for 12 weeks Route of administration: Oral Dosage form: Capsule
  Arms: Arm 3 - DehydraTECH-CBD in combination with DehydraTECH-semaglutide
Drug: Arm 4 - Rybelsus medication (semaglutide) alone — Normal clinical dose of 3.0 mg once daily for 4 weeks, ascending to 7.0 mg once daily for the remaining 8 weeks. Route of administration: Oral Dosage form: Capsule
  Arms: Arm 4 - Rybelsus medication (semaglutide) alone as a positive control.
Drug: Arm 5- Tirzepatide — Tirzepatide arm - 20mg for 4 weeks and then 40mg for 8 weeks
  Arms: Arm 5- DehydraTECH Tirzepatide

SUMMARY:
This is a Phase 1b, randomized, open-label, active-controlled, parallel, multiple-dose study comparing the safety, pharmacokinetics and efficacy of DehydraTECH Cannabidiol and Glucagon-like Peptide 1 (GLP-1) agonists alone and in combination, in overweight or obese, pre- and type 2 diabetic participants.

DETAILED DESCRIPTION:
The study duration is for a maximum study duration of 20 weeks and 6 days. All participants will be randomized to receive one of the 4 interventions- Arm 1- DehydraTECH-CBD alone; Arm2- DehydraTECH-semaglutide alone; Arm-3 DehydraTECH-CBD in combination with DehydraTECH-semaglutide or Arm 4 - Rybelsus medication (semaglutide) alone as a positive control. Arm 5- DehydraTECH Tirzepatide

Treatment period visits include safety assessments, including vital signs and physical examinations (symptom directed), as well as Patient reported outcome (PRO) questionnaires, body mass measures and a 15 to 20 mL blood sample.

ELIGIBILITY:
Inclusion criteria:

1. Clinically diagnosed as overweight or obese, with or without pre- or Type 2 diabetes with residual islet cell function.
2. For participants with pre- or Type 2 diabetes: diet controlled or receiving oral anti-diabetic treatment (metformin or other biguanides and/or sulphonylureas) who have received a stable dose for at least 3 months prior to enrollment.
3. Glycosylated haemoglobin levels of > 4.5 but ≤ 10%.
4. Have a BMI at Screening of ≥ 27.00 kg/m2 and ≤ 40 kg/m2 .
5. Willing to maintain a stable dose of oral anti-diabetic and/or lipid-lowering agents/medications that may have an effect on plasma glucose, insulin or lipid parameters for the duration of the study, where applicable.
6. No changes in diet for 4 weeks prior to randomisation (in the opinion of PI or designee), and willing to fast overnight prior to morning dosing during the course of the study. Willing to follow the recommendations for meals and water consumption around the time of each dose administration for the duration of the study (as defined in Section 7.3.3).
7. 18 to 65 years of age (inclusive at the time of informed consent).
8. Clinical laboratory values within normal range or as expected for the patient population or deemed not clinically significant (CS) by the PI or designee. One repeat test at Screening is acceptable for out-of-range CS values following approval by the PI or designee.
9. Estimated glomerular filtration rate (eGFR) within the normal range, using the 2021 CKD-EPI equation (> 60 mL / min / 1.73 m2).
10. Females must not be pregnant, planning pregnancy, or lactating, and must use acceptable, highly effective double contraception from Screening until 125 days after the last dose of IP administration. Effective forms of contraception are defined in Section 7.3.2. Females with same-sex partners (abstinence from penile-vaginal intercourse) or who are abstinent from heterosexual intercourse are not required to use contraception when this is their preferred and usual lifestyle. Women of childbearing potential (WOCBP) must have a negative pregnancy test at Screening and Day 1 and be willing to have additional pregnancy tests as required throughout the study. Women not of childbearing potential must be postmenopausal for ≥12 months (postmenopausal status is to be confirmed through testing of follicle stimulating hormone (FSH) levels ≥ 40 IU/L at Screening for amenorrhoeic female participants). Females must not donate ova from the first dose of IP until at least 125 days after the last dose of IP.
11. Males must be surgically sterile (> 30 days since vasectomy with no viable sperm), or if engaged in sexual relations with a WOCBP, either his partner must be surgically sterile (eg, tubal ligation, tubal occlusion, hysterectomy, bilateral salpingectomy, bilateral oophorectomy), or an acceptable, highly effective contraceptive method (see Section 7.3.2) must be used from Screening until study completion, including the Follow-up period. Males with same-sex partners (abstinence from penile-vaginal intercourse) or are abstinent from heterosexual intercourse are not required to use contraception when this is their preferred and usual lifestyle. Males must not donate sperm from the first dose of IP until at least 125 days after the last dose of IP.
12. Able and willing to attend the necessary visits to the study site and undertake all assessments.
13. Able and willing to provide written informed consent after the nature of the study has been explained and prior to the commencement of any study procedures.

Exclusion Criteria

A participant who meets any of the following exclusion criteria must be excluded from the study:

1. Personal or family history of medullary thyroid carcinoma (MTC) or multiple endocrine neoplasia type 2 (MEN2).
2. Participants with a history of, or currently undergoing treatment for, a thyroid disorder. Participants may still be eligible if they have an additional test confirming that TSH levels are within the normal range (at the discretion of the PI).
3. Participant is taking insulin (ie, they are insulin-dependent).
4. Taking the following categories of medicines: fibrates, Thiazolidinediones, therapeutic Omega-3 fatty acids (more than 4000 mg/day), alpha-glucosidase inhibitors and unwilling to abstain 2 weeks prior to dosing and for the duration of the study.
5. Currently taking a lipid lowering agent and a stable dose has not been maintained for at least 4 weeks prior to randomisation.
6. Use of anti-obesity medication within 90 days before enrollment.
7. Currently receiving a prohibited medication (Section 7.3.1) and unwilling to stop at the Screening visit and for the duration of the study.
8. Currently using an anti-hypertensive, with the exception of anti-hypertensives that are not relevant CYP450 inhibitors/inducers (listed in Table 2).
9. Medications that are not on a stable dose, directly prohibited per the protocol and mentioned in IBs as posing a risk for causing Drug-Drug-Interactions (DDIs) taken without the Investigator's review and approval. However, in case of concerns, the Investigator should consult with the Medical Monitor.
10. Vaccination with a live vaccine within 2 weeks prior to the first administration of IP.
11. Exposure to any significantly immune suppressing drug (including experimental therapies as part of a clinical study) within 4 months prior to Screening or 5-half lives, whichever is longer.
12. Use of any IP or investigational medical device within 30 days prior to Screening, or 5 half lives of the product (whichever is the longest) or participation in more than 4 investigational drug studies within 1 year prior to Screening.
13. Currently using or has used recreational cannabis, medicinal cannabis, cannabinoid medications (including Sativex®), or synthetic cannabinoid based medications within 30 days prior to study entry and unwilling to abstain for the duration for the study.
14. Current smoker, including cannabis user, and must not have used any tobacco or cannabis products within 30 days prior to Screening and unwilling to abstain for the duration for the study.
15. Positive toxicology screening panel (urine test including qualitative identification of barbiturates, tetrahydrocannabinol [THC], amphetamines, benzodiazepines, opiates, and cocaine), or alcohol breath test, except where a participant has a prescription and diagnosis (eg. ADHD on dexamphetamine, or opioids following an operation, etc.).
16. Known or suspected history of substance abuse or dependency or history of recreational intravenous (IV) drug use over the last 5 years (by self-declaration).
17. Regular alcohol consumption defined as > 10 standard drinks per week (where 1 standard drink = 360 mL of beer, 45 mL of 40% spirit or a 150 mL glass of wine) or > 4 standard drinks on any single day. Participant is unwilling to abstain from alcohol beginning 48 hours prior to Screening, the first administration of IP, and each subsequent visit.
18. A history of chronic pancreatitis, and/or acute pancreatitis within 180 days before randomisation.
19. Previous surgical obesity treatment (Cosmetic Surgery e.g. Liposuction allowed).
20. Any known or suspected history of epilepsy or recurrent seizures.
21. Diagnosis of a depressive disorder, regardless of severity, if antidepressants are currently being taken or have been used within 3 months prior to randomization. Exceptions include the use of antidepressants for non-depressive disorders (e.g., anxiety), provided a stable dose is maintained during the study. A diagnosis of depression without the use of antidepressants is not exclusionary.
22. Participant who has significant history of anxiety, suicidal ideation or self-harm and had to be institutionalised, or who appears to be unstable, in the opinion of the PI or designee.
23. Clinically significant cardiac, renal or hepatic impairment in the opinion of the PI or designee. For hepatic impairment, specifically excluding participants who have moderate (Child-Pugh B) or severe (Child-Pugh C) liver disease.
24. Genetic dyslipidemic condition in the opinion of the PI or designee.
25. Participants who would otherwise be eligible by BMI, but by subjective visual assessment are considered likely to have high muscle and low fat body composition (eg, body builders or strength sport athletes) in the opinion of the PI or designee.
26. Body weight > 150 kg..
27. Any abnormalities identified during the physical exam that in the opinion of the PI or designee, would prevent the participant from safe participation in the study.
28. Blood donation or significant blood loss within 60 days prior to the first administration of IP, or plasma donation within 7 days prior to the first administration of IP, and/or unwilling to abstain from donation of blood during the study.
29. History of severe allergic or anaphylactic reactions that in the opinion of the PI or designee might prevent the participant from safely participating in the study, or sensitivity to the IP or its constituents.
30. History of malignancy, unless cured more than 5 years prior to Screening (non-melanoma skin cancer excised more than 2 years prior to Screening, and cervical intraepithelial neoplasia that has been successfully cured more than 5 years prior to Screening, are permissible).
31. History or presence of a condition associated with significant immunosuppression.
32. History of life-threatening infection (eg, meningitis) within the past 5 years which may indicate risk to the participant at the discretion of the Investigator.
33. Infections requiring parenteral antibiotics within 6 months prior to Screening.
34. Fever (body temperature > 38°C) or symptomatic viral or bacterial infection within 2 weeks prior to Screening.
35. Systolic blood pressure of <100 mmHg or ≥180 mmHg and/or diastolic blood pressure of <80 mmHg or ≥120 mmHg, which in the opinion of the PI or designee may pose undue risk to the subject, or symptomatic uncontrolled hypotension or hypertension in the opinion of the PI or designee.
36. Moderate to severe daytime somnolence or daytime sleep disorders (e.g., narcolepsy).
37. Abnormal ECG findings at Screening that are considered by the PI or designee to be clinically significant.
38. Alkaline phosphatase (ALP), aspartate aminotransferase (AST), and/or alanine aminotransferase (ALT) > 1.5 × upper limit of normal (ULN) at Screening. One repeat test at Screening is acceptable for out-of-range values following approval by the PI or designee.
39. Positive test for hepatitis C antibody (HCV), hepatitis B surface antigen (HBsAg), or human immunodeficiency virus (HIV) antibody at Screening.
40. Poor pill swallowing ability.
41. Unwilling to refrain from strenuous exercise (including weightlifting) from 24 hours prior to each visit to the study site until the end of each visit.
42. Travel outside the country of residence planned during the study.
43. Any other significant disease or disorder, physical or psychological, or surgery (within the past 3 months prior to Screening) which, in the opinion of PI or designee, may either put the participant at risk because of participation in the study, or may influence the result of the study, or the participant's ability to comply with the protocol or complete the study per protocol.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2024-12-04 (Actual); Primary Completion 2025-07-31 (Actual); Study Completion 2025-07-31 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment-emergent adverse events (TEAEs) and Serious adverse events | Baseline to Day 113 post first dose administration

SECONDARY OUTCOMES:
Number of participants with abnormal laboratory parameters from baseline to end of study (EOS) | Baseline to Day 113 post first dose administration
Number of participants who have a magnitude of decrease in HbA1c (1% or greater) and/or bodyweight (5% or greater) from baseline. | Baseline to Day 113 post first dose administration
Number of participants with change in fasting glucose from baseline | Baseline to Day 113 post first dose administration
Number of participants with change in insulin cholesterol levels from baseline | Baseline to Day 113 post first dose administration
Number of participants with change in inflammation (hsCRP)from baseline | Baseline to Day 113 post first dose administration
Number of participants with change in estimated glomerular filtration rate from baseline | Baseline to Day 113 post first dose administration
Number of participants with change in liver enzymes from baseline | Baseline to Day 113 post first dose administration

CONTACTS AND LOCATIONS:
Locations (7):
- Australia (7):
  - Paratus Clinical Pty Ltd, Blacktown Trial Clinic, Blacktown, New South Wales
  - Emeritus - Sydney, Botany, New South Wales
  - Canopy Clinical Sutherland, Miranda, New South Wales
  - Canopy Clinical Wollongong, Wollongong, New South Wales
  - Paratus Clinical Brisbane Pty Ltd, Herston, Queensland
  - CMAX Clinical Research, Adelaide, South Australia
  - Emeritus - Melbourne, Camberwell, Victoria

IPD SHARING:
Plan to Share IPD: No